CLINICAL TRIAL: NCT02077426
Title: Heart Failure and Regional Specific Exercise Training Stimulus
Acronym: HF-RSTS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00051711
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-03

CONDITIONS: Heart Failure; Sedentary
Keywords: Functional Capacity; Exercise Independence; Peripheral; Strength
MeSH Terms: conditions — Heart Failure; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regional Specific Training (RSTS) (Experimental): The RSTS protocol was designed to focus on specific peripheral muscle groups without imposing a significant cardiorespiratory strain. Each exercise involved contractions with moderate load but with an extended duration of up to six minutes. Eight specific exercises were performed to target all major muscle groups and enable the routine to be completed within 60 minutes including warm-up, rest periods and stretching between exercises, and cool down exercises
  Interventions: Other: Regional Specific Training (RSTS)

INTERVENTIONS:
Other: Regional Specific Training (RSTS) — The RSTS protocol was designed to focus on specific peripheral muscle groups without imposing a significant cardiorespiratory strain. Each exercise involved contractions with moderate load but with an extended duration of up to six minutes. Eight specific exercises were performed to target all major muscle groups and enable the routine to be completed within 60 minutes including warm-up, rest periods and stretching between exercises, and cool down exercises.

SUMMARY:
The aim of this study is to determine whether heart failure patients can tolerate a four-weeks of a new exercise training regimen that targets peripheral tissues (Regional Specific Training Stimulus-RSTS) and has been show to produce significant benefits in aerobic capacity and strength in healthy subjects aged 70+years who were at risk for losing functional independence.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 55 and 90
* Diagnosed with heart failure (NYHA class II-III)
* Receiving optimal medical therapy
* Sedentary (≤ 30 min/wk structured physical activity)
* Peak VO2 between 10 and 30 mL/kg/min.

Exclusion Criteria:

* Oxygen dependent
* Recent medications changes (within 3 months)
* Fixed-rate pacemakers
* Uncontrolled hypertension
* Type I diabetes
* Organ transplant
* Bariatric surgery
* Renal failure (stage 4 or 5)

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Subject Adherence & Compliance | 4 Weeks
  The number of training sessions attended and successfully completed divided by the total number of planned sessions
One Repetition Maximum (1RM) | 4 Weeks
  Skeletal muscle strength assessed using a one repetition maximum (1RM) measurement obtained for the seated row, chest press, leg press and handgrip.
Senior Fitness Test | 4 Weeks
  The Senior Fitness Test is a previously validated battery of 6 physical tasks of daily living used to assess strength, flexibility and endurance in order to detect and predict future limitations in functional capacity. The test is designed to evaluate physical fitness domains including upper-body strength (Arm Curl), lower-body strength (Chair Sit-Stand), upper and lower body flexibility (Back Scratch and Chair Sit and Reach), balance and coordination (8 foot Up and Go), and endurance (Six Minute Walk).

CONTACTS AND LOCATIONS:
Overall Officials: Jason D Allen, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Center for Living; Wallace Clinic, Durham, North Carolina, United States